CLINICAL TRIAL: NCT05102955
Title: Turkish Validity and Reliability of the Visual Function Classification System (VFCS) in Children With Cerebral Palsy (CP)
Brief Title: Turkish Validity and Reliability of the Visual Function Classification System (VFCS)
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, assistant professor, Kahramanmaras Sutcu Imam University
Other Study IDs: haticeadiguzel
Record Dates: First submitted 2021-10-15; First posted 2021-11-02 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy; Visual Impairment; Visual Disorder; Cerebral Visual Impairment; Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Visual Function Classification System (VFCS); validity; reliability; Visual Impairment; Visual Disorder
MeSH Terms: conditions — Cerebral Palsy; Vision Disorders; Blindness, Cortical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Observational Questionnaires: All one Group/ Visual Function Classification System(VFCS), Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), Communication Function Classification System(CFCS) Questionnaires will be assessed by the different raters(physiotherapists). But Visual Function Classification System(VFCS) will be assesed also by the parents.
  Interventions: Other: Observational questionnaires

INTERVENTIONS:
Other: Observational questionnaires — All one Group/ Visual Function Classification System(VFCS), Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), Communication Function Classification System(CFCS) Questionnaires will be assessed by the different raters (physiotherapists). But Visual Function Classification System(VFCS) will be assesed also by the parents.
  Other Names: Assessments

SUMMARY:
Cerebral Palsy (CP) is the most common childhood disorder that occurs with a lesion in the developing infant brain, seen in 2-3/1000 live births. CP is a posture, movement and tone disorder that occurs due to prenatal or postnatal causes. It is not progressive, but since the anatomy of the lesion and the physical development of the individual are not completed, the course of the disorder may vary throughout life. Accompanied by motor dysfunctions, it varies according to clinical types. In addition to this, various visual, sensory and behavioral problems, speech disorders that cause learning difficulties and cognitive problems can also be observed. Ophthalmic disorders are the most common problem in CP and can also affect the developmental process of the patient. Since ophthalmic disorders and neurological deficits are associated in CP, the relationship between neurological disorder and ophthalmic disorders has been investigated in the literature. The aim of this study is to establish the Turkish validity and reliability of the Visual Function Classification System (VFCS) specific to individuals with Cerebral Palsy (CP).

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common childhood disorder that occurs with a lesion in the developing infant brain, seen in 2-3/1000 live births. CP is a posture, movement and tone disorder that occurs due to prenatal or postnatal causes. It is not progressive, but since the anatomy of the lesion and the physical development of the individual are not completed, the course of the disorder may vary throughout life. Accompanied by motor dysfunctions, it varies according to clinical types. In addition to this, various visual, sensory and behavioral problems, speech disorders that cause learning difficulties and cognitive problems can also be observed. Ophthalmic disorders are the most common problem in CP and can also affect the developmental process of the patient. Since ophthalmic disorders and neurological deficits are associated in CP, the relationship between neurological disorder and ophthalmic disorders has been investigated in the literature. Studies show that 60-70% of children with CP also have CVI. CVI is defined as a lack of visual function resulting from damage or disruption of the retrogeniculate visual pathways (optic radiations, occipital cortex, visual associative areas) in the absence of any major ocular disease. This involvement of the retrogeniculate visual pathways is common in CP, given that the lesions most commonly underlying this condition also affect the visual areas of the brain. CVI is defined as bilateral loss of central visual function (visual acuity) caused by neurological damage to the visual cortex and⁄or visual pathway structures. It is most commonly caused by hypoxic ischemia causing periventricular leukomalacia (PVL) in the preterm infant. Disturbance of the oculomotor system is also typical in CP. Abnormalities in functions such as fixation, tracking and saccadic movements; Strabismus and abnormal ocular movements are also frequently described. With the participation of visual relational areas, visual perception and integration disorders, which are often seen as visual cognitive disorders, can occur when the child reaches school age. These impairments should be investigated even when visual functions such as visual acuity and visual field are normal or mildly impaired.Gross Motor Classification System (GMFCS) and Manual Skill Classification System (MACS) are used by clinicians to obtain a clear picture of how motor skills of individuals with CP, mobility levels in daily life and independence levels of hand functions are affected. However, although it is known that children with CP have visual effects, the methods in which visual functions are classified are insufficient. Therefore, Baranello et al. A tool has been developed to classify the visual function classification system. The aim of this study is to establish the Turkish validity and reliability of the Visual Function Classification System (VFCS) specific to individuals with Cerebral Palsy (CP).

ELIGIBILITY:
Inclusion Criteria:

-Children with CP diagnosed with CP between the ages of 1-18 with visual perception problems and visual impairments

Exclusion Criteria:

* Individuals with CP whose parents did not sign the voluntary consent form

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with CP of different clinical types in the 1-18 age range
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Function Classification System (VFCS) | The same physiotherapists and parents (P) of children with CP will re-apply the VFCS classifications to individuals with CP up to 15-day after the first assessment.
  The VFCS was developed empirically following a step-by step process to classify visual abilities of children with CP in everyday life. VFCS levels will be scored as; LEVEL I: Uses visual function easily and successfully in vision-related activities. LEVEL II: Uses visual function successfully but needs self-initiated compensatory strategies. LEVEL III: Uses visual function but needs some adaptations. LEVEL IV: Uses visual function in very adapted environments but performs just part of vision-related activities. LEVEL V: Does not use visual function even in very adapted environments.The same TWO physiotherapists and parents (M) of children with CP will re-apply the VFCS classifications to individuals with CP at 15-day intervals.

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | Day 1
  Gross Motor Function Classification System (GMFCS), which defines both disease severity and disease course, is used to classify motor impairment in children with cerebral palsy. This system is a system that is used to inform the family about the instant performance of the child. Gross Motor Function Classification System is a valid and reliable standardized system that classifies the gross motor functions of children with CP between the ages of 0-12 at five levels. Children with cerebral palsy are least dependent at level 1 and most dependent at level 5 in motor functions.
Manual Ability Classification System (MACS) | Day 1
  MACS determines how children with CP use their hands while holding objects in daily activities. MACS; defines five levels. The determination of levels is based on the child's ability to hold objects to himself and the need for assistance and adaptation in performing manual activities in daily life. MACS aims to categorize what a child does in general, not how well he performs during a specific test. MACS assesses the usual general ability to hold objects, not the function of the two hands separately or their ability to grasp. Instead of considering the difference in function between the two hands, MACS considers how the child handles objects appropriate for his age. MACS can be used for children aged 4-18. Levels I, II, III include children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
Communication Function Classification System (CFCS) | Day 1
  The CFCS assesses the communication functions of an individual with CP in daily life on a five-level scale. The differences between the five levels of the CFCS are based on important aspects of functional communication, namely the performance of the sender and receiver roles, the speed of the conversation, and the communication partner type. Turkish validity and reliability were established.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adiguzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Hatice Adıgüzel, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adiguzel Tat H, Karadeniz PG, Apaydin U, Efkere PA, Ergun N, Elbasan B. Reliability and Cross-Cultural Validation of the Turkish Version of the Visual Function Classification System (VFCS) for Children with Cerebral Palsy. Dev Neurorehabil. 2024 Nov;27(8):328-336. doi: 10.1080/17518423.2024.2413133. Epub 2024 Oct 13. PMID 39396187